CLINICAL TRIAL: NCT03607890
Title: Phase 2 Study of Nivolumab and Relatlimab in Advanced Mismatch Repair Deficient Cancers Resistant to Prior PD-(L)1 Inhibitor
Brief Title: Study of Nivolumab and Relatlimab in Advanced Mismatch Repair Deficient Cancers Resistant to Prior PD-(L)1 Inhibitor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J18102; IRB00173534 (Other: JHMI IRB); P50CA062924 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Refractory MSI - H Solid Tumors Prior of PD-(L) 1 Therapy; MSI-H Tumors
Keywords: Relatlimab; Nivolumab; Immunotherapy; Anti - PD-1; Anti - LAG-3; Antibodies; MSI; MMR deficient; Microsatellite instability
MeSH Terms: conditions — Turcot syndrome; Microsatellite Instability | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Nivolumab and Relatlimab (Experimental): 480mg/160mg (co-administered)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- Cohort 2: Nivolumab and Relatlimab (Experimental): 480mg/960mg or 480mg/160mg (sequential administration)
  Interventions: Drug: Nivolumab; Drug: Relatlimab
- Cohort 3: Nivolumab and Relatlimab (Experimental): 480mg/480mg (sequential administration)
  Interventions: Drug: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Patients will receive treatment every 28 days for up to 2 years. Nivolumab will be administered IV on day 1 (28 day cycle).
  Other Names: anti-PD-1, OPDIVO
  Arms: Cohort 1: Nivolumab and Relatlimab
Drug: Relatlimab — Patients will receive treatment every 28 days up to 2 years. Relatlimab will be administered IV on day 1 (28 day cycle).
  Other Names: BMS-986016
  Arms: Cohort 1: Nivolumab and Relatlimab
Drug: Nivolumab — Patients will receive treatment every 28 days for up to 2 years. Nivolumab will be administered IV on day 1 (28 day cycle).
  Other Names: anti-PD-1, OPDIVO
  Arms: Cohort 2: Nivolumab and Relatlimab
Drug: Relatlimab — Patients will receive treatment every 28 days up to 2 years. Relatlimab will be administered IV on day 1 (28 day cycle).
  Other Names: BMS-986016
  Arms: Cohort 2: Nivolumab and Relatlimab
Drug: Nivolumab — Patients will receive treatment every 28 days for up to 2 years. Nivolumab will be administered IV on day 1 (28 day cycle).
  Other Names: anti-PD-1, OPDIVO
  Arms: Cohort 3: Nivolumab and Relatlimab
Drug: Relatlimab — Patients will receive treatment every 28 days up to 2 years. Relatlimab will be administered IV on day 1 (28 day cycle).
  Other Names: BMS-986016
  Arms: Cohort 3: Nivolumab and Relatlimab

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of nivolumab and relatlimab in patients with microsatellite instability high (MSI-H) solid tumors refractory to prior PD-(L)1 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Have metastatic or locally advanced mismatch repair deficient/MSI-H disease.
* Patients must have received prior PD-1/PD-L1 inhibitor therapy
* Patients with the presence of at least one measurable lesion.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study - specified laboratory tests.
* Documented left ventricular ejection fraction (LVEF) ≥ 50% - 6 month prior to drug administration.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Known history or evidence of brain metastases.
* Require any antineoplastic therapy.
* History of prior treatment with anti-LAG3.
* Had chemotherapy, radiation, or steroids within 14 days prior to study treatment.
* Had any investigational cytotoxic drug within 4 weeks prior to study treatment.
* Have received any investigational drugs, a live vaccine, any allergen hyposensitization therapy, growth factors or major surgery within 28 days prior to study treatment.
* Major surgery
* Hypersensitivity reaction to any monoclonal antibody.
* Has an active known or suspected autoimmune disease.
* Has a diagnosis of immunodeficiency.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* Requires daily supplemental oxygen
* History of interstitial lung disease.
* Significant heart disease
* History of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Infection with HIV or hepatitis B or C at screening.
* Has an active infection.
* Unable to have blood drawn.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior life-threatening toxicity to anti-PD-1, anti-PD-L1, anti-PD-L2,or anti-CTLA4
* Woman who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | 4 years

SECONDARY OUTCOMES:
Number of participants experiencing study drug-related toxicities | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided